CLINICAL TRIAL: NCT05628610
Title: Tislelizumab Combined With Chemotherapy or Radiotherapy in the Treatment of Advanced or Recurrent Metastatic Elderly Esophageal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tisle-001
Record Dates: First submitted 2022-11-18; First posted 2022-11-28 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — tislelizumab; Radiation; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tislelizumab combined with radiotherapy (Experimental)
  Interventions: Drug: Tislelizumab; Radiation: Radiation
- Tislelizumab combined with chemotherapy (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Paclitaxel; Drug: Platinum: cisplatin, carboplatin, naidaplatin and other platinum drugs

INTERVENTIONS:
Drug: Tislelizumab — 200mg d1, Q3W
Radiation: Radiation — Radiotherapy dose: 5,000 c G y / 30f
  Arms: Tislelizumab combined with radiotherapy
Drug: Paclitaxel — Paclitaxel: 150mg / m2 ,d1, q3w
  Arms: Tislelizumab combined with chemotherapy
Drug: Platinum: cisplatin, carboplatin, naidaplatin and other platinum drugs — cisplatin, carboplatin, naidaplatin and other platinum drugs
  Arms: Tislelizumab combined with chemotherapy

SUMMARY:
To compare the objective response rate (ORR) and safety of tislelizumab combined with chemotherapy and Tislelizumab combined with radiotherapy in elderly patients with esophageal cancer with advanced or recurrent metastasis

ELIGIBILITY:
Inclusion Criteria:

* Signed a written informed consent and volunteered to join the study;
* Patients with esophageal squamous cell carcinoma confirmed by pathological histological and / or immunohistochemical examination or progressing after surgical resection, (the 8th edition, 2017) with UICC / AJCC TNM stage cT4N0-2M0, c any TN3M0, or c any T any NM1 (clinical stage IV);
* Unresectable advanced, recurrent, or metastatic oesophageal SCC;
* Age: 70 years old;
* E CO G P S 0-2
* Has not received any systemic antitumor treatment for esophageal cancer, including radiotherapy, chemotherapy, targeted, immunotherapy, etc.;
* At least one measurable lesion was present
* Main organs have normal function, including:

A) Routine blood tests (no blood components, cell growth factors, whitening agents, platelets, anemia drugs are allowed within 14 days before the first use of the study drug) Leukocyte count was at 3.0109/L Neutrophil count was at 1.0109/L Platelet count was at 8,0109/L Hemoglobin was at 80 g / L b) Blood biochemical examination: Total bilirubin was at 1.5 ULN ALT ≤ 2.5×ULN ，AST ≤2.5×ULN ， Serum creatinine of 1.5 ULN, or creatinine clearance of 45 mL/min (Cocheroft-Gault formula, see Annex 2)

-The subjects had good compliance and cooperated with the follow-up

Exclusion Criteria:

* There is uncontrollable pleural effusion, pericardial effusion or ascites that requires repeated drainage;
* Poor nutritional status, BMI <18.5 Kg / m2; if corrected after symptomatic nutritional support, further enrollment can be considered after evaluation by the principal investigator;
* Gastrointestinal bleeding (bleeding volume> 200ml / day);
* Patients adjudged by the researchers to have deep ulcers;
* Previous history of allergy to monoclonal antibodies, any component of tirellizumab, paclitaxel, cisplatin, or other platinum drugs;
* Has received or are receiving any of the following treatments:

A) Any radiotherapy, chemotherapy, or other antitumor drugs directed against the tumor; Study drug b) Treatment with immunosuppressive drugs or systemic hormones for immunosuppression purposes within 2 weeks of the first study drug (dose or equivalent dose> 10mg / day); inhaled or topical steroids and doses> 10mg / day prednisone or equivalent dose of adrenal corticoid replacement in the absence of active autoimmune disease; The c) Acceptance of a live attenuated vaccine within 4 weeks before the first use of the study drug; d) Major surgery or severe trauma within 4 weeks prior to the first use of the study drug;

* History of any active autoimmune or autoimmune disease, including but not limited to: interstitial pneumonia, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (considered after HRT); patients with psoriasis or asthma / allergy in childhood remission and adults without any intervention, but patients requiring bronchodilator are not included;
* A history of immunodeficiency, including positive HIV testing, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation or allogeneic bone marrow transplantation;
* Poor clinical cardiac symptoms or disease, including but not limited to:

Such as (1) heart failure of grade NYHAII or above; (2) unstable angina pectoris; (3) myocardial infarction within 1 year; (4) clinical significance of supraventricular or ventricular arrhythmia without clinical intervention or clinical intervention is not well controlled;

* Severe infection (CTCAE> 2) within 4 weeks before initial use of study drug, such as severe pneumonia, bacteremia, or infection complications requiring hospitalization; baseline chest imaging indicates active lung inflammation, symptoms or signs of infection within 14 days prior to initial use of study drug, or requiring oral or intravenous antibiotics, except for prophylactic antibiotics;
* Patients with active tuberculosis infection by medical history or CT examination, or active tuberculosis infection within 1 year prior to enrollment, or active tuberculosis infection within 1 year before enrollment, or before enrollment but without formal treatment;
* The presence of active hepatitis B (HBV DNA 2000 IU / mL or 104 copies / mL), hepatitis C (hepatitis C antibody positive, and HCV RNA above the lower limit of the analysis method);
* According to the investigator, there are other factors present that may lead to the forced termination of the study, such as other serious illness (including mental illness) requiring combined treatment, alcohol abuse, substance abuse, family or social factors, that may affect the safety or compliance of the subject.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 12 months
  Clinical response of treatment according to RESIST v1.1 criteria (ORR, objective response rate).

SECONDARY OUTCOMES:
progression free survival | 12 months
  The length of time from enrollment until the time of progression of disease (PFS, progression-free survival).

IPD SHARING:
Plan to Share IPD: No